CLINICAL TRIAL: NCT06580054
Title: Pembrolizumab for Orbital and Periocular Cutaneous Squamous Cell Carcinoma (cSCC)
Brief Title: Pembrolizumab for the Treatment of Locally Advanced and/or Recurrent Orbital or Periocular Cutaneous Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2021.025; NCI-2024-06539 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00229341 (Other: University of Michigan Comprehensive Cancer Center); UMCC 2021.025 (Other: University of Michigan Comprehensive Cancer Center)
Record Dates: First submitted 2024-08-18; First posted 2024-08-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Cutaneous Squamous Cell Carcinoma of the Head and Neck; Recurrent Cutaneous Squamous Cell Carcinoma of the Head and Neck; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8
MeSH Terms: interventions — Magnetic Resonance Spectroscopy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI or CT and photographs of tumor throughout the study.
  Interventions: Procedure: Computed Tomography; Other: Digital Photography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Other: Digital Photography — Undergo photographs of tumor
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; QL2107; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with orbital (eye socket) and/or periorbital (surrounding the eye socket) cutaneous squamous cell cancer (cSCC) that has spread to nearby tissue or lymph nodes (locally advanced) or has come back after a period of improvement (recurrent). Skin cancers that are close to the eye or on the eyelid often have more genetic (heredity) changes than other types of cancers. This means that the deoxyribonucleic acid (DNA) (the building blocks of the body that determine such things as the color of the hair) in tumor tissue has been altered compared to normal tissue. It is thought cancer cells with these DNA changes are more likely to respond to a type of drug called immunotherapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Pembrolizumab is approved for patients with recurrent or metastatic cSCC not amenable (responsive) to cure by surgery or radiation. Giving pembrolizumab may work better in treating patients with locally advanced or recurrent orbital and/or periorbital cSCC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether treatment of patients with locally advanced or recurrent orbital and/or periocular cSCC with pembrolizumab will be associated with tumor response.

SECONDARY OBJECTIVES:

I. To assess the globe preservation rate among patients with locally advanced or recurrent orbital and/or periocular cSCC treated with pembrolizumab.

II. To determine whether treatment with pembrolizumab of patients with locally advanced or recurrent orbital and/or periocular cSCC will prevent progression of disease.

EXPLORATORY OBJECTIVES:

I. To evaluate next generation sequencing (NGS) and correlate with response to therapy for patients with available tissue.

II. Correlate visual function to location and size of tumor over the course of treatment.

III. To identify if the presence of human papillomavirus (HPV) in the cSCC affects the tumor response.

IV. To determine the duration of response (DOR) at 2 years.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo magnetic resonance imaging (MRI) or computed tomography (CT) and photographs of tumor throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 9 weeks for 52 weeks and then every 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent.
* Histologically confirmed diagnosis of locally advanced or diffuse or recurrent orbital or periorbital cutaneous squamous cell carcinoma.
* Female participants:

  * A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) as defined.
    * A WOCBP who agrees to follow the contraception guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* The participant provides written informed consent for the trial.
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Absolute neutrophil count (ANC) ≥ 1500/uL.
* Platelets ≥ 100000/uL.
* Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L.

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* Creatinine ≤ 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) ≥ 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN.

  * Creatinine clearance (CrCl) should be calculated per institutional standard.
* Total bilirubin ≤ 1.5 x ULN OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 x ULN.
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 x ULN (≤ 5 x ULN for participants with liver metastases).
* International normalized ratio (INR) OR prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.
* Have recovered from toxicities and/or complications from any prior major surgery before starting study treatment.
* Have a life expectancy of at least 12 weeks.
* Patients with human immunodeficiency virus (HIV) adequately controlled on antiretroviral therapy.
* Patients with known hepatitis B infection (defined as hepatitis B surface antigen [HbsAg] reactive) should be on suppressive anti hepatitis B virus (HBV) therapy, and patients with history of hepatitis C infection (defined as hepatitis C virus [HCV] ribonucleic acid [RNA] detected) must complete curative antiviral treatment with HCV viral load below limit of quantification. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.

Exclusion Criteria:

* Has any other histologic type of skin cancer other than invasive squamous cell carcinoma as the primary disease under study.
* A WOCBP who has a positive pregnancy test within 72 hours prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a negative serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to enrollment. Participants must have recovered from all adverse events (AEs) due to previous therapies to ≤ grade 1 or baseline. Participants with ≤ grade 2 neuropathy may be eligible.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist [registered trademark]) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an interventional investigational device within 4 weeks prior to the first dose of study intervention. Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years. The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers like ocular surface squamous cell neoplasia.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
* Has severe hypersensitivity (≥ grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of active tuberculosis (TB) (bacillus tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue (e.g., hematopoietic stem cell transplant [HSCT])/solid organ transplant.
* Has a history of any of the following cardiovascular conditions:

  * Myocardial infarction within 6 months of enrollment.
  * Active unstable angina.
  * Congestive heart failure (≥ New York Heart Association Classification Class II)
  * Cerebral vascular accident/stroke within 6 months of enrollment.
  * Serious cardiac arrhythmia requiring medication. The classification of "serious" is at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Up to 2 years
  Will be calculated from the tumor partial and complete responses based on immune-related Response Evaluation Criteria In Solid Tumors. Will be reported with exact 95% binomial confidence intervals.

SECONDARY OUTCOMES:
Globe preservation | Up to 2 years
  To assess the globe preservation rate among patients. External and slit lamp photography will be obtained during the Ophthalmic exams
Time to progression | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Worden, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No